CLINICAL TRIAL: NCT01569815
Title: An Open Label, Parallel-group Study to Determine Multiple Dose Pharmacokinetics of LCZ696 and Its Metabolites in Subjects With Mild and Moderate Renal Impairment Compared to Matched Healthy Subjects With Normal Renal Function
Brief Title: Pharmacokinetics of LCZ696 in Subjects With Mild and Moderate Renal Impairment Compared to Healthy Subjects With Normal Renal Function
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CLCZ696A2204; 2007-005480-96 (EudraCT Number)
Record Dates: First submitted 2012-03-30; First posted 2012-04-03 (Estimated); Results first posted 2015-08-27 (Estimated); Last update posted 2015-10-19 (Estimated); Status verified 2015-09

CONDITIONS: Mild and Moderate Renal Impairment
Keywords: Renal Impairment,; LCZ696
MeSH Terms: conditions — Lymphoma, Follicular; Renal Insufficiency | interventions — sacubitril and valsartan sodium hydrate drug combination

ARMS (1):
- LCZ696 400 mg (Experimental): LCZ696 400 mg once daily for 5 days
  Interventions: Drug: LCZ696

INTERVENTIONS:
Drug: LCZ696 — LCZ696 400 mg once daily

SUMMARY:
The purpose of this study is to determine the multiple dose pharmacokinetics of LCZ696 and its metabolites in subjects with mild to moderate renal impairment and to evaluate the safety of LCZ696 in this population.

ELIGIBILITY:
Inclusion Criteria:

1. Male, and female subjects of non-child bearing potential,
2. Subjects were to weigh at least 50 kg to participate in the study,
3. and body mass index < 40 kg/m2
4. Subjects were able to communicate well with the investigator, to understand and comply with the requirements of the study;
5. Subjects were able to understand and sign the written informed consent;

For renal insufficient subjects:

1. stable renal disease without evidence of renal progressive

   * mild renal function: calculated CrCl of 50-≤80 mL/min
   * moderate renal function: calculated CrCl of 30-<50 mL/min
2. Vital signs:

   * oral body temperature between 35.0-37.8 °C
   * systolic blood pressure, 95-180 mm Hg
   * diastolic blood pressure, 60-110 mm Hg
   * pulse rate, 54-95 bpm

For healthy subjects only

1. A serum creatinine with a calculated CrCl of >80 mL/min
2. Vital signs:

   * oral body temperature between 35.0-37.2 °C
   * systolic blood pressure, 95-140 mm Hg
   * diastolic blood pressure, 60-100 mm Hg
   * pulse rate, 45-90 bpm

Exclusion Criteria:

1. Current use of ACE inhibitors, valsartan, and drugs that were known as CYP2C9 substrates, potassium-sparing diuretics;
2. Smokers;
3. History of renal transplant at any time in the past and on immunosuppressant therapy;
4. Dialysis patients;
5. Medical history of clinically significant ECG abnormalities or a family history of a prolonged QT-interval syndrome;
6. Any surgical or medical condition which may significantly alter the absorption, distribution, metabolism or excretion of any drug substance; Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2009-02; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (3):
- Novartis Investigative Site, Neuss, Germany
- Novartis Investigative Site, Moscow, Russia
- Novartis Investigative Site, Belgrade, Serbia

RESULTS

PARTICIPANT FLOW:
Groups:
- Mild Renal Impaired; Mild Renal Impaired Matched Healthy Subjects; Moderate Renal Impaired Subjects; Moderate Renal Impaired Matched Healthy Subjects: LCZ696 400 mg once daily for 5 days
Period: Overall Study
Arm/Group | Mild Renal Impaired | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Started | 8 | 8 | 8 | 8
Completed | 8 | 8 | 8 | 8
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Mild Renal Impaired Subjects; Mild Renal Impaired Matched Healthy Subjects; Moderate Renal Impaired Subjects; Moderate Renal Impaired Matched Healthy Subjects: LCZ696 400 mg once daily for 5 days
- Total: Total of all reporting groups
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects | Total
Number analyzed (Participants) | 8 | 8 | 8 | 8 | 32
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.0 (10.88) | 50.6 (11.70) | 54.5 (8.33) | 53.9 (8.95) | 52.5 (9.72)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 3 | 3 | 8
  Male | 7 | 7 | 5 | 5 | 24
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0 | 0
  White | 8 | 8 | 8 | 8 | 32
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Time to Reach Maximum Peak Plasma Concentration (Tmax) After Single Dose (Day 1), and After Multiple Dose Administration (Day 5)
Description: Blood samples will be collected for the determination of plasma concentrations of VAL489 (valsartan), AHU377( Sacubitril) and LBQ657 (a human metabolite of sacubitril)
Time Frame: Day 1 and day 5
Measure: Median (Full Range); unit: hr
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 8
hr
  AHU377 day 1, single dose of LCZ696 400 mg | 1 [0.5 to 2.0] | 0.5 [0.5 to 1.0] | 0.5 [0.5 to 4.0] | 0.5 [0 to 2]
  AHU377 day 5, multiple doses of LCZ696 400 mg Q.D. | 1 [0.5 to 2.0] | 0.5 [0.0 to 2.0] | 0.5 [0.5 to 1.0] | 0.5 [0.5 to 1.0]
  LBQ657 day 1, single dose of LCZ696 400 mg | 3 [2 to 4] | 2 [2 to 3] | 3 [2 to 8] | 3 [2 to 3]
  LBQ657 day 5, multiple doses of LCZ696 400 mg Q.D. | 3 [2 to 4] | 3 [2 to 3] | 3 [2 to 4] | 3 [2 to 4]
  VAL489 day 1, single dose of LCZ696 400 mg | 2.5 [2 to 3] | 2 [2 to 4] | 2 [1 to 6] | 2 [1 to 3]
  VAL489 day 5,multiple doses LCZ696 400 mg Q.D. | 2.5 [1 to 4] | 2 [1 to 3] | 2 [2 to 2] | 2 [2 to 2]

2. Primary Outcome: Maximum Peak Plasma Concentration (Cmax) Observed After Single Dose (Day 1), and After Multiple Dose Administration (Day 5)
Description: as for outcome 1
Time Frame: Day 1, day 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng/mL
  AHU377 day 1, single dose of LCZ696 400 mg | 4220 (1514) | 3995 (1368) | 3539 (1414) | 3743 (1486)
  AHU377 day 5, multiple doses of LCZ696 400 mg Q.D | 3904 (1780) | 3125 (1729) | 4109 (1739) | 3756 (1644)
  LBQ657 day 1, single dose of LCZ696 400 mg | 17575 (3500) | 15200 (2958) | 18175 (3210) | 16000 (2451)
  LBQ657 day 5, multiple doses of LCZ696 400 mg Q.D. | 27150 (6449) | 16838 (3063) | 28988 (7861) | 18375 (3215)
  VAL489 day 1, single dose of LCZ696 400 mg | 7208 (3606) | 6215 (1588) | 6178 (2584) | 7981 (2059)
  VAL489 day 5,multiple dose LCZ696 400 mg Q.D. | 6873 (4348) | 6275 (2242) | 7665 (2612) | 8006 (3895)

3. Primary Outcome: Area Under the Concentration-time Curve (AUC0-24) From Time Zero to 24- Hour Post-dose (Day 1), and After Multiple Dose Administration (Day 5)
Description: as for outcome 1
Time Frame: Day 1 and day 5
Population: FAS
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 8
ng*hr/mL
  AHU377 day 1, single dose of LCZ696 400 mg | 5679 (1864) | 5396 (1197) | 5359 (2287) | 5963 (2559)
  AHU377 day 5, multiple doses of LCZ696 400 mg Q.D | 5656 (1859) | 5221 (1162) | 5283 (2267) | 5716 (1849)
  LBQ657 day 1, single dose of LCZ696 400 mg | 226159 (49810) | 144500 (15533) | 262422 (52115) | 154871 (31504)
  LBQ657 day 5, multiple dose of LCZ696 400 mg Q.D. | 371331 (99259) | 172335 (21925) | 437134 (146930) | 190598 (44468)
  VAL489 day 1, single dose of LCZ696 400 mg | 62411 (43846) | 40658 (11401) | 47135 (21560) | 50220 (19732)
  VAL489 day 5,multiple dose LCZ696 400 mg Q.D | 59223 (50669) | 39517 (17227) | 51777 (18967) | 56460 (31412)

4. Primary Outcome: Elimination Half-life (t1/2) After Multiple Dose (Day 5) Administration
Description: as for outcome 1
Time Frame: Day 5
Population: FAS
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 8
hr
  AHU377 day 5, multiple doses of LCZ696 400 mg Q.D | 1.6 (0.6) | 4.7 (6.0) | 2.9 (2.3) | 1.8 (1.2)
  LBQ657 day 5, multiple dose of LCZ696 400 mg Q.D | 21.1 (8.3) | 12.6 (1.7) | 23.7 (5.0) | 12.3 (2.2)
  VAL489 day 5,multiple dose LCZ696 400 mg Q.D | 15.4 (4.7) | 14.5 (3.7) | 22.7 (14.6) | 12.4 (3.0)

5. Primary Outcome: Systemic Clearance From Plasma Following Extravascular Administration (CL/F) After Multiple Dose Administration (Day 5)
Description: as for outcome 1
Time Frame: Day 5
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 8
mL/hr
  AHU377 day 5, multiple doses of LCZ696 400 mg Q.D | 38261 (14002) | 39137 (10451) | 42704 (17238) | 37902 (14487)
  LBQ657 day 5, multiple dose of LCZ696 400 mg Q.D | NA (NA) — LBQ657 is a metabolite of AHU377, and hence LBQ657 CL/F values are not relevant. | NA (NA) — LBQ657 is a metabolite of AHU377, and hence LBQ657 CL/F values are not relevant. | NA (NA) — LBQ657 is a metabolite of AHU377, and hence LBQ657 CL/F values are not relevant. | NA (NA) — LBQ657 is a metabolite of AHU377, and hence LBQ657 CL/F values are not relevant.
  VAL489 day 5,multiple dose LCZ696 400 mg Q.D | 4636 (17080) | 6499 (3876) | 4929 (3260) | 5988 (6568)

6. Primary Outcome: Accumulation Ratio (Racc) After Multiple Dose Administration (Day 5)
Description: as for outcome 1
Time Frame: Day 5
Population: FAS
Measure: Mean (Standard Deviation); unit: Ratio (AUC0-24, day 5)/(AUC0-24, day 1)
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 8
Ratio (AUC0-24, day 5)/(AUC0-24, day 1)
  AHU377 day 5, multiple dose of LCZ696 400 mg Q.D | 1.0 (0.1) | 1.0 (0.2) | 1.0 (0.2) | 1.0 (0.2)
  LBQ657 day 5, multiple dose of LCZ696 400 mg Q.D | 1.64 (0.27) | 1.19 (0.09) | 1.6 (0.3) | 1.2 (0.1)
  VAL489 day 5,multiple dose LCZ696 400 mg Q.D | 1.0 (0.4) | 0.9 (0.2) | 1.3 (0.6) | 1.1 (0.5)

7. Primary Outcome: Renal Clearance From Plasma (CLr) After Multiple Dose Administration (Day 5)
Description: as for outcome 1
Time Frame: Day 5
Population: FAS
Measure: Mean (Standard Deviation); unit: mL/hr
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 8
mL/hr
  AHU377 day 5,multiple dose of LCZ696 400 mg Q.D | 81.2 (30.5) | 129.1 (97.0) | 48.9 (36.3) | 143.9 (145.2)
  LBQ657 day 5, multiple dose of LCZ696 400 mg Q.D | 253.1 (99.0) | 499.0 (251.3) | 111.0 (81.4) | 486.0 (85.7)
  VAL489 day 5,multiple dose LCZ696 400 mg Q.D | 141.6 (84.7) | 313.8 (144.5) | 73.2 (43.1) | 317.0 (109.0)

8. Primary Outcome: Amount of Drug Excreted Into the Urine From Time Zero to 24-hours Post-dose (Ae0-24) After Single Dose (Day 1), and After Multiple Dose Administration (Day 5)
Description: as for outcome 1
Time Frame: Day 1 and Day 5
Measure: Mean (Standard Deviation); unit: ug
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 8
ug
  AHU377 day 1, single dose of LCZ696 400 mg | 360.2 (99.1) | 1560 (1294) | 419.4 (351.1) | 2083 (2496)
  AHU377 day 5, multiple dose of LCZ696 400 mg Q.D | 426.2 (120.3) | 734.5 (662.8) | 316.8 (362.9) | 790.8 (872.6)
  LBQ657 day 1, single dose of LCZ696 400 mg | 52687 (17107) | 68397 (17535) | 29653 (11767) | 75699 (15612)
  LBQ657 day 5, multiple dose of LCZ696 400 mg Q.D | 87768 (21278) | 83254 (35800) | 43952 (20678) | 92113 (22572)
  VAL489 day 1, single dose of LCZ696 400 mg | 7206 (3082) | 13792 (5250) | 4156 (2634) | 16902 (4628)
  VAL489 day 5,multiple dose LCZ696 400 mg Q.D | 6849 (3852) | 11625 (6186) | 3713 (1843) | 16385 (8260)

9. Secondary Outcome: Change in Mean 24-hours Sodium Clearance From Baseline to Day 7
Description: Sodium clearance will be measured in urine from baseline until Day 7
Time Frame: From baseline to Day 7
Population: FAS
Measure: Mean (Standard Deviation); unit: mmol/day
Arm/Group | Mild Renal Impaired Subjects | Mild Renal Impaired Matched Healthy Subjects | Moderate Renal Impaired Subjects | Moderate Renal Impaired Matched Healthy Subjects
Number analyzed (Participants) | 8 | 8 | 8 | 8
mmol/day
  Baseline | 107.13 (51.709) | 150.25 (50.349) | 110.65 (40.169) | 158.38 (56.835)
  Day 1 | 143.24 (36.293) | 185.75 (38.592) | 129.26 (36.510) | 196.13 (51.99)
  Day 2 | 118.4 (48.036) | 134.88 (46.603) | 95.63 (37.799) | 134.38 (38.774)
  Day 3 | 117.38 (51.798) | 127.50 (56.488) | 97.89 (29.745) | 141.00 (43.808)
  Day 4 | 140.70 (52.127) | 133.38 (60.656) | 107.38 (43.007) | 142.88 (40.470)
  Day 5 | 161.68 (80.545) | 133.50 (53.596) | 104.45 (34.775) | 178.00 (44.156)
  Day 6 | 163.32 (13.81) | 129.38 (65.600) | 106.42 (25.427) | 184.25 (81.310)
  Day 7 | 141.63 (72.63) | 117.50 (48.794) | 102.02 (45.256) | 146.25 (69.405)

ADVERSE EVENTS:
Groups:
- LCZ696 400 mg - Mild - Renal Impaired Patients: LCZ696 400 mg - Mild - Renal impaired patients
- LCZ696 400 mg - Mild - Matched Healthy Subjects: LCZ696 400 mg - Mild - Matched healthy subjects
- LCZ696 400 mg - Moderate - Renal Impaired Patients: LCZ696 400 mg - Moderate - Renal impaired patients
- LCZ696 400 mg - Moderate - Matched Healthy Subjects: LCZ696 400 mg - Moderate - Matched healthy subjects
- LCZ696 400 mg - All Healthy Subjects: LCZ696 400 mg - All healthy subjects
Arm/Group | LCZ696 400 mg - Mild - Renal Impaired Patients | LCZ696 400 mg - Mild - Matched Healthy Subjects | LCZ696 400 mg - Moderate - Renal Impaired Patients | LCZ696 400 mg - Moderate - Matched Healthy Subjects | LCZ696 400 mg - All Healthy Subjects
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/8 | 0/8 | 0/8 | 0/16
Other Adverse Events (participants affected / at risk) | 7/8 | 3/8 | 8/8 | 1/8 | 4/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | LCZ696 400 mg - Mild - Renal Impaired Patients (N=8) | LCZ696 400 mg - Mild - Matched Healthy Subjects (N=8) | LCZ696 400 mg - Moderate - Renal Impaired Patients (N=8) | LCZ696 400 mg - Moderate - Matched Healthy Subjects (N=8) | LCZ696 400 mg - All Healthy Subjects (N=16)
Postural orthostatic tachycardia syndrome (Cardiac disorders) | 2 | 0 | 2 | 0 | 0
Sinus bradycardia (Cardiac disorders) | 1 | 0 | 4 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 1
Fatigue (General disorders) | 0 | 1 | 0 | 0 | 1
Hyperkalaemia (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0 | 0
Somnolence (Nervous system disorders) | 0 | 1 | 0 | 0 | 1
Haematuria (Renal and urinary disorders) | 1 | 0 | 1 | 0 | 0
Leukocyturia (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 1 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 0
Diastolic hypertension (Vascular disorders) | 1 | 0 | 0 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 1 | 0 | 0
Hypotension (Vascular disorders) | 1 | 0 | 0 | 1 | 1
Orthostatic hypertension (Vascular disorders) | 2 | 0 | 2 | 0 | 0
Orthostatic hypotension (Vascular disorders) | 2 | 2 | 5 | 1 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial